CLINICAL TRIAL: NCT04941404
Title: A Single Arm, Open-label, Multicenter, Phase Ib Study of TQ05105 Tablets in Subjects With aGVHD
Brief Title: A Study of TQ05105 Tablets in Subjects With Glucocorticoid-Refractory Acute Graft-Versus-Host Disease (aGVHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-Ib-01
Record Dates: First submitted 2021-06-22; First posted 2021-06-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Glucocorticoid-Refractory aGVHD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ05105 tablets (Experimental): Participants began oral administration of TQ05105 tablets at 10 mg twice daily (BID),followed by 5 mg or 15 mg BID depending on the situation of the study. twice daily in 28-day cycle until disease progression/intolerance occurs or the sponsor terminates the study.
  Interventions: Drug: TQ05105 tablets

INTERVENTIONS:
Drug: TQ05105 tablets — Participants began oral administration of TQ05105 tablets at 10 mg twice daily (BID),followed by 5 mg or 15 mg BID depending on the situation of the study. twice daily in 28-day cycle until disease progression/intolerance occurs or the sponsor terminates the study.

SUMMARY:
This is an open-label,single arm,Phase Ib study,in order to evaluate the safety,tolerability, preliminary efficacy and pharmacokinetics of TQ05105 tablets in subjects with Glucocorticoid-Refractory aGVHD

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participated in the study and signed an informed consent, with good compliance.
2. Aged 12-75, gender is not limited.
3. Subjects who has received allogeneic hematopoietic stem cell transplantation (allo-HSCT) previously.
4. Clinically suspected grades II to IV acute GVHD as per MAGIC guidelines.
5. Drug resistance after glucocorticoid treatment.
6. Absolute neutrophils count (ANC) >1×109/L,Platelet(PLT)≥20×109/L within 48 hours before initial treatment.
7. Male or female subjects should agree use an adequate method of contraception during the study and within 6 months after the end of the study (such as intrauterine devices , contraceptives or condoms) ;No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

Exclusion Criteria:

1. Subjects with a history of progressive multifocal leukoencephalopathy.
2. Subjects with many factors influencing oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction, etc.).
3. Arteriovenous thrombotic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, etc..
4. Severe respiratory diseases (requiring mechanical ventilation or O2 saturation < 90%), active tuberculosis, pulmonary hypertension and pulmonary embolism, etc..
5. Subjects with a history of psychotropic drug abuse and can not quit or have mental disorders.
6. Subjects with any severe and/or uncontrolled disease, including:

(1) Unsatisfactory blood pressure control with more than 2 drugs (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥ 100mmHg) ; (2) Patients with grade ≥2 myocardial ischemia or infarction, arrhythmias (including QTc≥480ms), and grade ≥2 congestive heart failure (New York Heart Association classification); (3) Uncontrolled active infections including bacteria, fungi, parasites or viruses such ascytomegalovirus, Epstein-Barr virus, and human herpes virus 6; (4) Cirrhosis, active hepatitis; (5) Human immunodeficiency virus(HIV) positive, active syphilis; (6) Creatinine clearance rate < 30 mL/min,calculated by Cockcroft Gault formula; (7) Patients with epilepsy and need treatment. 7. Subjects with evidence of recurrence of primary disease or relapsed after allo-HSCT treatment.

8. There were grade 2 or higher toxicity (except aGVHD) caused by previous allo HSCT treatment.

9. Subjects who received allo-HSCT more than once in the past. 10. Subjects who received more than one kind of systemic treatment for Glucocorticoid-Refractory aGVHD.

11. The clinical manifestations were new-onset chronic GVHD or overlapping GVHD syndrome with both acute and chronic GVHD features.

12. Allergic to the investigational drug or its ingredients. 13. Subjects who used Janus kinase inhibitor (JAK) therapy after receiving Allo-HSCT.

14. Subjects who participated in other clinical trials within 4 weeks before initial administration.

15. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the subjects or affect the completion of the study, or subjects who are considered unsuitable for other reasons.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Drug tolerance of the first cycle (Stage 1) | Day 28 after initial administration
  Dose-limiting toxicity events related to the investigational drug occured within 28 days after initial administration
Objective Response Rate (ORR) at Day 28 (Stage 2) | Day 28 after initial administration
  Percentage of subjects with complete response (CR) or very good partial response (VGPR) or partial response (PR) at Day 28

SECONDARY OUTCOMES:
CR Rate at Day 28 | Day 28 after initial administration
  Percentage of subjects with CR at Day 28
ORR at Day 28 and Day 56 | Day 28 and Day 56 after initial administration
  Percentage of subjects with CR or VGPR or PR at Day 28 and Day 56
Duration of Response (DOR) | From initial administration to day 30 after the last administration
  From date of first recorded remission to date of first recorded disease progression or date of starting any new systemic therapy for aGVHD
Cumulative dose of glucocorticoid at Day 56 | Day 56 after initial administration
  Totally and weekly cumulative dose of glucocorticoid of each subject,from initial administration to Day 56 or the day end of therapy
Event Free Survival (EFS） | From initial administration to Day 30 day after the last administration
  From the date of initial administration to the date of recurrence/progression of hematological diseases or transplant failure or death from any cause
Overall Survival (OS) | From initial administration to day 30 days after the last administration
  Time from randomization to death
Incidence of Malignancy Relapse/Progression(MR),Non-Relapse Mortality(NRM) | From initial administration to 30 days after the last administration
  From the date of first administration to the date of death due to recurrence/progression of non hematological diseases; the date of recurrence or progression of hematological diseases
Incidence of adverse events (AEs) and serious adverse events (SAEs) | From initial administration to day 30 after the last administration
  Incidence of AEs and SAEs
Tmax | 7 days after initial administration
  The pharmacokinetic parameters were measured after single and multiple administration: peak time(Tmax)
Cmax | 7 days after initial administration
  The pharmacokinetic parameters were measured after single and multiple administration: peak concentration(Cmax)
AUC0-t | 7 days after initial administration
  The pharmacokinetic parameters were measured after single and multiple administration: area under the blood concentration-time curve (AUC0-t)

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Hematology Hospital of the chinese Academy of Medical Sciences, Tianjing, Tianjing
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang